CLINICAL TRIAL: NCT04055480
Title: A Multi-centre, Randomised, Two-period, Crossover Study to Evaluate Home Use of Closed-loop Applying Faster Insulin Aspart Versus Standard Insulin Aspart
Brief Title: Closing the Loop in Adults With Type 1 Diabetes Under Free Living Conditions
Acronym: AP@Home04_P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Insel Gruppe AG, University Hospital Bern (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor of Metabolic Technology, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136248_APHome04
Record Dates: First submitted 2019-08-06; First posted 2019-08-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes
Keywords: closed-loop; artificial pancreas; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop using standard rapid-acting insulin (Active Comparator): Unsupervised home use of day and night hybrid closed loop insulin delivery system (CamAPS FX) for 8 weeks using standard rapid-acting insulin
  The CamAPS FX closed-loop system comprises
  Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) An Android smartphone hosting CamAPS FX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system to monitor CGM/insulin data.
  Interventions: Device: Closed-loop using standard rapid-acting insulin
- Closed-loop using faster insulin aspart (Experimental): Unsupervised home use of day and night hybrid closed loop insulin delivery system (CamAPS FX) for 8 weeks using faster insulin aspart
  The CamAPS FX closed-loop system comprises
  Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) An Android smartphone hosting CamAPS FX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system to monitor CGM/insulin data.
  Interventions: Device: Closed-loop using faster insulin aspart

INTERVENTIONS:
Device: Closed-loop using standard rapid-acting insulin — Closed-loop using standard rapid-acting insulin
  Arms: Closed-loop using standard rapid-acting insulin
Device: Closed-loop using faster insulin aspart — Closed-loop using faster insulin aspart
  Arms: Closed-loop using faster insulin aspart

SUMMARY:
The main objective of this study is to determine whether home use of day and night closed loop insulin delivery under free living conditions applying faster insulin aspart (FiAsp) is non-inferior to home use of closed-loop applying standard insulin aspart.

This is a double-blind, multi-centre, randomised, crossover design study, involving a run-in period followed by two study periods during which glucose levels will be controlled either by an automated closed-loop system using standard rapid acting insulin analogue or by an automated closed-loop system using faster insulin aspart in random order.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. Subjects will have regular contact with the study team during the home study phase including 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM during home stay. Secondary outcomes are the HbA1c, time spent with glucose levels above and below target, as recorded by CGM, and other CGM based metrics.

DETAILED DESCRIPTION:
Purpose of clinical trial The purpose is to determine whether home use of day and night closed loop applying faster insulin aspart is not inferior to home use of closed loop applying standard insulin aspart.

Study objectives The study objective is to compare day and night automated closed-loop glucose control using faster acting insulin aspart with closed loop control using standard insulin aspart.

1. EFFICACY: The objective is to assess the efficacy of day and night automated closed-loop glucose control applying standard rapid-acting insulin analogue in maintaining CGM glucose levels within the target range from 3.9 to 10.0 mmol/l, as compared to day and night closed-loop using faster acting insulin aspart
2. SAFETY: The objective is to evaluate the safety of day and night automated closed-loop glucose control in terms of episodes of severe hypoglycaemia, hyperglycaemia and other adverse events and adverse device effects.
3. UTILITY: The objective is to determine the percentage of time when closed-loop was operational, and usability and acceptance of the closed-loop system.

Study Design A double-blind, multi-centre, randomised, two-period crossover study, contrasting day and night automated closed-loop glucose control applying standard rapid acting insulin analogue with day and night closed-loop control applying faster acting insulin aspart.

Study Efficacy Endpoints The primary outcome is the time spent in the target glucose range from 3.9 to 10.0 mmol/l based on CGM glucose levels during the free living phase.

Secondary outcomes include time spent above and below the target glucose range, based on CGM levels.

Safety Evaluation Frequency of severe hypoglycaemic episodes as defined by American Diabetes Association, frequency of severe hyperglycaemia (>20 mmol/l) and / or significant ketosis (plasma ketones >3mmol/l) and nature and severity of other adverse events.

Utility Evaluation Percentage of time spent in closed-loop. Usability and acceptance of the closed-loop system will be assessed using a patient experience questionnaire at the end of the second intervention. Additionally, human factor questionnaires will be administered following recruitment and at the end of each intervention arm.

Sample Size 24 adults completing the study. Up to 30 subjects will be recruited to allow for dropouts.

Maximum duration of study for a subject 20 weeks (5 months)

Recruitment The subjects will be recruited through the adult diabetes outpatient clinics or other established methods at participating centres.

Consent Participants will be asked to provide written informed consent.

Baseline Assessment Eligible subjects will undergo a baseline evaluation including a blood sample for the measurement of HbA1c, renal, liver functions, full blood count, thyroid functions and coeliac antibody screen (if not done in the previous 3 months). Urine pregnancy test will be done in females. Additional centre specific assessments will also be undertaken. Human factor questionnaires will be administered.

Study Training and Run-in Period Training sessions on the use of study CGM, insulin pump and closed-loop system will be provided by the research team. During the 2-4 weeks run-in period, subjects will use study CGM and insulin pump and will have regular contact with the research team. At the end of the run-in period, for compliance and to assess the ability of the subject to use the CGM and study pump safely, before the start of the first home study phase, at least 7 days of CGM data need to be recorded and safe use of study insulin pump demonstrated. CGM and insulin pump data during the run-in period will be used to assess baseline glucose control and optimise treatment before the start of the first home study phase.

Competency Assessment Competency on the use of study insulin pump, study CGM and closed-loop system will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required.

Randomisation Eligible subjects will be randomised using randomisation software to the use of closed-loop with faster acting aspart or to closed-loop with standard insulin aspart.

Automated closed-loop Training on the use of closed-loop will be provided by the research team. Automated closed-loop control will be commenced and during the 2-3 hour training the participant will operate the system under the supervision of the clinical team. Competency on the use of closed-loop system will be evaluated. Subjects will be advised to use automated closed-loop system for next 8 weeks

Cross-over Assessment At the end of the first intervention human factor questionnaires will be administered.

There will be no washout period in phase 3 extension.

End of study assessments A patient experience questionnaire will be given at the end of the second intervention. Additionally human factor questionnaires will be administered.

Procedures for safety monitoring during trial Standard operating procedures for monitoring and reporting of all adverse events and adverse device events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

Subjects will be asked to test and record blood ketones if their finger-stick glucose is above 14 mmol/l as part of the safety assessment for hyperglycaemia.

A data monitoring and ethics committee (DMEC) will be informed of all serious adverse events and any unanticipated adverse device/method effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of patients on safety grounds

A subject may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

* Serious adverse events
* Significant protocol violation or noncompliance
* Failure to satisfy competency assessment
* Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest
* Pregnancy, planned pregnancy, or breast feeding
* Allergic reaction to insulin
* Technical grounds (e.g. subject relocates)

ELIGIBILITY:
Inclusion Criteria:

1. The subject has type 1 diabetes as defined by WHO
2. The subject is 18 years of age or older
3. The subject will have been on an insulin pump for at least 6 months with good knowledge of insulin self-adjustment including carbohydrate counting
4. The subject is treated with one of the rapid acting or ultra-rapid acting insulin analogues (Insulin Aspart, faster acting insulin Aspart, Insulin Lispro or Insulin Glulisine)
5. HbA1c <10% (86mmol/mol) for phase 3, based on analysis from central laboratory or equivalent
6. The subject is willing to perform regular finger-prick blood glucose monitoring, with at least 2 measurements per day
7. The subject is willing to wear closed-loop system at home and at work place
8. The subject is willing to follow study specific instructions including the use of bolus calculator for all meals / snacks
9. The subject is willing to upload pump and CGM data at regular intervals
10. Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening.

Exclusion Criteria:

1. Non-type 1 diabetes mellitus
2. Subjects who are living alone
3. Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
4. Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
5. Known or suspected allergy against insulin or previous reaction to FiAsp
6. Subjects with clinically significant nephropathy (eGFR < 45ml/min), neuropathy or active retinopathy (defined as presence of maculopathy or more than background diabetic retinopathy changes) as judged by the investigator
7. More than one episode of severe hypoglycaemia as defined by American Diabetes Association (42) in preceding 12 months (Severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions including episodes of hypoglycaemia severe enough to cause unconsciousness, seizures or attendance at hospital.)
8. Total daily insulin dose > 2 IU/kg/day
9. Subject is pregnant or breast feeding or planning pregnancy within next 10 months
10. Severe visual impairment
11. Severe hearing impairment
12. Lack of reliable telephone facility for contact
13. Subject not proficient in English (UK), French (Switzerland) or German (Germany, Switzerland and Austria)

Additional exclusion criteria specific for Austria

1. Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
2. Positive alcohol breath test.
3. Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 antibodies, anti-HIV2 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM). | 8 week intervention period

SECONDARY OUTCOMES:
Time spent above target glucose (3.9 to 10.0 mmol/l) based on continuous subcutaneous glucose monitoring (CGM) | 8 week intervention period
Time spent below target glucose (3.9 to 10.0 mmol/l) based on continuous subcutaneous glucose monitoring (CGM) | 8 week intervention period
Average, standard deviation and coefficient of variation of glucose levels based on continuous subcutaneous glucose monitoring | 8 week intervention period
The time with glucose levels < 3.5 mmol/l <3.0mmol/l and <2.8 mmol/l based on continuous subcutaneous glucose monitoring | 8 week intervention period
The time with glucose levels in the significant hyperglycaemia, as based on continuous subcutaneous glucose monitoring (glucose levels > 16.7 mmol/l) | 8 week intervention period
Low Blood Glucose Index (LBGI) based on continuous subcutaneous glucose monitoring | 8 week intervention period
Total, basal and bolus insulin dose | 8 week intervention period

OTHER OUTCOMES:
Safety evaluation will comprise the number of episodes of hypoglycaemia, significant ketonemia (>3.0mmol/l) as well as nature and severity of any other adverse events. | Through study completion, an average of 5 months
Utility evaluation is the frequency and duration of use of the closed-loop system at home. | 8 week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, Principal Investigator — University of Cambridge
Locations (4):
- Medical University of Graz, Graz, Austria
- Inselspital, Bern University Hospital, Bern, Switzerland
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.

REFERENCES:
- [Derived] Haliloglu B, Boughton CK, Lakshman R, Ware J, Nwokolo M, Thabit H, Mader JK, Bally L, Leelarathna L, Wilinska ME, Allen JM, Hartnell S, Evans ML, Hovorka R. Postprandial Glucose Excursions with Ultra-Rapid Insulin Analogs in Hybrid Closed-Loop Therapy for Adults with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jul;26(7):449-456. doi: 10.1089/dia.2023.0509. Epub 2024 Feb 27. PMID 38315506